CLINICAL TRIAL: NCT01837992
Title: Evaluation of Safety and Efficacy of Two Primaquine Dosing Regimens for the Radical Treatment of Plasmodium Vivax Malaria in Vanuatu and Solomon Islands
Brief Title: Safety and Efficacy of Primaquine for P. Vivax
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Menzies School of Health Research (Other)
Collaborators: Walter and Eliza Hall Institute of Medical Research (Other); Ministry of Health, Vanuatu (Other Government); Ministry of Health, Solomon Islands (Other Government); World Health Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VanSI_2013
Record Dates: First submitted 2013-03-25; First posted 2013-04-23 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard dose (Active Comparator): Participants will receive a standard 3-day treatment course of artemether-lumefantrine at the standard age-based dosage, and will be administered the standard recommended primaquine dose of 0.25mg/kg for 14 consecutive days.
  Interventions: Drug: Primaquine
- High dose (Active Comparator): Participants will receive a standard 3-day treatment course of artemether-lumefantrine at the standard age-based dosage, and will be administered a primaquine dose of 0.5mg/kg/day for 14 consecutive days.
  Interventions: Drug: Primaquine
- Control (Other): Participants will receive a standard 3-day treatment course of artemether-lumefantrine at the standard age-based dosage, but will not receive primaquine until the time of confirmed recurrent parasitaemia or completion of 3 months follow up.
  Interventions: Drug: delayed primaquine

INTERVENTIONS:
Drug: Primaquine
  Arms: High dose; Standard dose
Drug: delayed primaquine
  Arms: Control

SUMMARY:
The Melanesian states of the Western Pacific (Papua New Guinea, Solomon Islands and Vanuatu) represent a unique and especially prescient challenge to malaria control and elimination.

While the use of bed nets and other vector control and case management measures have achieved major advances in overall malaria control, the P. vivax and P. ovale species account for an ever-increasing burden of clinical disease.

The lack of effective treatment of the hypnozoite stages of infection with these species result in ongoing relapses and a continuing reservoir of infection.

The only known drug effective for treatment of the hypnozoite stage is primaquine; however the safe and effective dose of this drug in malaria treatment is still unclear.

A recent study evaluated the safety and efficacy of two primaquine dosing regimens (0.25mg/kg and 0.5mg/kg) in a population in New Ireland province, PNG. This study aims to replicate this methodology in Vanuatu and Solomon Islands, to provide a more complete picture of primaquine efficacy and safety in each of the three countries of this region.

DETAILED DESCRIPTION:
Study Aims

Primary To define and compare the efficacy of standard (0.25mg/kg/day for 14 days) and high-dose (0.5mg/kg/day for 14 days) primaquine in preventing early relapses from P. vivax in Solomon Islands and Vanuatu.

Secondary To measure safety and toxicity of primaquine when administered as a standard or high-dose regimen in Melanesian adults and children in Solomon Islands and Vanuatu.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12 months to 60 years
2. Melanesian background and living in local area
3. Microscopically (based on field microscopy) or RDT confirmed P.vivax regardless of parasite density. Mixed infections (P.falciparum-P.vivax and P.malariae-P.vivax) can be included.

Exclusion Criteria:

1. Any signs of severe malaria (see WHO definitions) including: impaired consciousness, respiratory distress, severe anaemia (Hb<5), multiple seizures, frequent vomiting/ inability to swallow tablets, prostration, jaundice, hypotension, abnormal bleeding or hypoglycaemia.
2. Clinical evidence of non-malarial illness (such as pneumonia or otitis media)
3. Severe malnutrition (weight-for-age nutritional Z score [WAZ] <60th percentile)
4. Permanent disability, which prevents or impedes study participation.
5. Treatment with primaquine in the previous 14 days
6. Residence or planned travel outside the study area during the follow-up period (precluding supervised treatment and follow-up procedures)
7. Known or suspected pregnancy
8. Currently breastfeeding
9. A positive rapid test for G6PD deficiency (Binax or Carestart RDT)

Following later PCR-based confirmation of malaria speciation, there may be some post-hoc exclusion of subjects in whom it is thought the initial field-based microscopic diagnosis may have been incorrect.

Ages: 12 Months to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Numbers of Plasmodium vivax relapses per person-years of follow- | 12 months
  Total number of microscopically diagnosed (including both symptomatic and asymptomatic infections), PCR-confirmed relapses with Plasmodium vivax in participants in each treatment arm over the 3-month follow-up period, expressed as number of relapses per person-years of follow-up.

SECONDARY OUTCOMES:
Safety and toxicity (1): Numbers with mild adverse events | 12 months
  Numbers in each treatment arm experiencing any documented adverse event defined as "mild" (not severe enough to interfere with daily activities).
Safety and toxicity (2) Numbers with moderate adverse events | 12 months
  Numbers in each treatment arm experiencing any documented adverse event defined as "moderate" (severe enough to interfere with daily activities but not severe enough to warrant admission to hospital).
Safety and toxicity (3) Numbers with severe adverse events | 12 months
  Numbers in each treatment arm experiencing any documented adverse event defined as "severe" (severe to warrant admission to hospital or to be considered a risk for death or disability arising from the event).
Safety and toxicity (4) Numbers with any adverse events | 12 months
  Numbers in each treatment arm experiencing any documented event (defined as either mild, moderate or severe as above).
Safety and toxicity (5) Numbers with assumed significant haemolysis | 12 months
  Numbers in each treatment arm experiencing any of the following:
  1. Haemoglobinuria on dipstick examination
  2. Scleral icterus
  3. Haemoglobin concentration fall by more than 25% of baseline or absolute concentration <5g/dL
Safety and toxicity (6) Numbers with significant methaemoglobinaemia | 12 months
  Numbers in each treatment arm experiencing any of the following:
  1. Cyanosis (blue tongue, lips and peripheries)
  2. Measured methaemoglobin saturation (using Masimo Rad-57 plus oximeter) >15%
  3. Measured oxygen saturation <85%

CONTACTS AND LOCATIONS:
Locations (4):
- Solomon Islands (2):
  - Tetere Hospital, Guadalcanal Province, Honiara, Guadalcanal Province
  - Aoki Hospital, Malaita Province, Auki, Malaita Province
- Vanuatu (2):
  - Northern Provincial Hospital, Nambauk Aid Post, V.F.H.A Dispensary and Fanafo Dispensary, Luganville, Sanma
  - Toroa Dispensary, NTM Health Centre and Vila Central Hospital, Port Vila, Shefa Province